CLINICAL TRIAL: NCT03714607
Title: Management of Vaginal Prolapse Using Laser Therapy: Randomized Controlled Trial
Brief Title: Laser Therapy in Managing Vaginal Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Themos Grigoriadis, Assistant Professor, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 310/26-04-2018
Record Dates: First submitted 2018-10-13; First posted 2018-10-22 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Cystocele; Vaginal Vault Prolapse; Rectocele; Enterocele
MeSH Terms: conditions — Cystocele; Pelvic Organ Prolapse; Rectocele; Hernia | interventions — Lasers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser (Experimental): Erbium Yttrium Aluminum Garnet (Er:YAG) laser therapies
  Interventions: Device: Erbium Yttrium Aluminum Garnet (Er:YAG) laser
- Control (No Intervention): No intervention

INTERVENTIONS:
Device: Erbium Yttrium Aluminum Garnet (Er:YAG) laser — 5 Er:YAG laser therapies vaginally administered at monthly intervals
  Other Names: Fotona
  Arms: Laser

SUMMARY:
Efficacy of laser therapy in postmenopausal women with symptomatic prolapse stage >1. Assessment tools will include prolapse stage quantification system (POP-Q) and validated condition related questionnaires.

DETAILED DESCRIPTION:
Postmenopausal women with symptomatic cystocele and/or rectocele stage 2 or 3 will be 1:1 randomly allocated to Er:YAG laser or watchful waiting group. Participants in the Er:YAG laser group will receive laser therapies at monthly intervals, while participants in the watchful waiting group will receive no treatment. All outcomes in both groups will be evaluated at baseline, 4-months and 6-months from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic prolapse stage >1 (cystocele, vaginal vault prolapse, enterocele, rectocele) according to POP-Q System
* Negative Pap-smear

Exclusion Criteria:

* Asymptomatic prolapse
* prolapse stage <=1
* prolapse of uterus
* presence of any type of genital infections (i.e herpes, vaginitis etc)
* vaginal bleeding
* underlying pathologies that could interfere in patients compliance (i.e psychiatric)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 30 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Quantification System (POP-Q) | Change from baseline to 4-6 months
  Physical examination

SECONDARY OUTCOMES:
Pelvic Floor Distress Inventory Short Form (PFDI) | Change from baseline το 4-6 months
  Total score is calculated by adding the scores of 3 scales (Urogenital Distress Inventory (UDI)-6, Pelvic Organ Prolapse Distress Inventory (POPDI)-6 and Colorectal Anal Distress Inventory (CRADI)-8) with a possible range from 0 to 300. Each scale-item could receive values from 0 to 4 applying to a score ranging from 0 to 100 for each scale. The higher the score the more intense are the symptoms.
International Consultation on Incontinence Modular Questionnaire-Female Lower Urinary Tract Symptoms (ICIQ-FLUTS) | Change from baseline to 4-6 months
  It is a 12-items questionnaire evaluating nocturia, urgency, bladder pain, frequency, hesitancy, straining, intermittency, urinary incontinence (UI) (urge, stress and unexplained), frequency of urinary incontinence and nocturnal enuresis. Filling, voiding and incontinence symptoms subscales range from 0 to 15, 0 to 12 and 0 to 20, respectively. Additionally, it evaluates impact of individual symptoms with bothering scales that are not incorporated in the overall scores.
Pelvic Floor Impact Questionnaire short Form | Change from baseline to 4-6 months
  Includes 3 domains (incontinence impact questionnaire (IIQ), Pelvic Organ Prolapse Impact Questionnaire (POPIQ) and Colorectal-anal Impact Questionnaire (CRAIQ) with overall 21-items (7 items in each domain). The total score of PFIQ-7 ranges from 0 to 300 (each domain may receive scores from 0 to 100). The highest the score the greater is the impact
Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire Short form | Change from baseline to 4-6 months
  It includes 12 items corresponding to behavioral-emotive, physical and partner related domains. Likert scale ranging from always (0 score) to never (4 score) is encompassed. Scores are obtained for all domains individually. The sum of all scores create a total PISQ score. PISQ total score range from 0-125. Higher values indicate better sexual functioning.
Patients Global Impression of Improvement | 4-6 months
  It is a single-item questionnaire aiming to evaluate patients impression of improvement following therapeutic intervention.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 3 months post-treatment
  Women will be asked to keep a diary reporting any adverse events occuring.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Athanasiou, Associate Proffesor, Study Director — National and Kapodistrian University of Athens, Greece
Locations (1):
- Urogynecological Unit of Alexandra Hospital, Athens, Greece

REFERENCES:
- [Derived] Athanasiou S, Pitsouni E, Cardozo L, Zacharakis D, Petrakis E, Loutradis D, Grigoriadis T. Can pelvic organ prolapse in postmenopausal women be treated with laser therapy? Climacteric. 2021 Feb;24(1):101-106. doi: 10.1080/13697137.2020.1789092. Epub 2020 Jul 28. PMID 32720552